CLINICAL TRIAL: NCT07151378
Title: Intestinal Levodopa + Entacapone Therapy (Lecigon®) to Counteract Dopaminergic Desensitization and Neuropsychiatric Complications in Parkinson's Disease
Acronym: INITIATE-LECIG
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2025-521048-39-00; 2025-521048-39-00 (EU CTIS Number)
Record Dates: First submitted 2025-06-27; First posted 2025-09-03 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: PARKINSON DISEASE (Disorder)
Keywords: LECIG; device assisted therapy; motor and non-motor fluctuations; dopaminergic complications; impulse control disorder; levodopa seeking; dopamine dysregulation syndrom; dopamine agonist; intestinal levodopa
MeSH Terms: conditions — Parkinson Disease; Disruptive, Impulse Control, and Conduct Disorders | interventions — Levodopa; Carbidopa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best oral medical treatment: the patients in this arm will be continue the treatment they were in f (Active Comparator): Amog others L_DOPA + Decarboxymethylasehemmer Dopamine agonist Amantadine COMT-Inhibitors
  Interventions: Drug: Best oral medication
- Lecigon® (Experimental)
  Interventions: Drug: LECIG (levodopa, carbidopa, entacapone intestinal gel)

INTERVENTIONS:
Drug: LECIG (levodopa, carbidopa, entacapone intestinal gel) — intestinal L-Dopa + entacapone (Lecigon®)
  Arms: Lecigon®
Drug: Best oral medication — Best oral medication
  Arms: Best oral medical treatment: the patients in this arm will be continue the treatment they were in f

SUMMARY:
This study is a Phase III multicentric randomized controlled trial with parallel group design and waiting list in patients that have an indication to undergo intestinal L-Dopa + entacapone (Lecigon®) under the existing indication criteria (according to SmPC (Fachinformation) Lecigon®). As primary endpoint, we will analyze the difference of the pre-interventional baseline and 6-month follow-up on the "hyperdopaminergic symptoms" corresponding to section 3 of the "Ardouin Behavioural Scale" hypothesizing on the superiority of LECIG therapy compared to best medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent document prior to any study related assessments/procedures. 2. Able to adhere to the study visit schedule and other protocol requirements. 3. Female Subject of childbearing potential1 and male subjects with female partner of childbearing potential1 is willing to use highly effective contraceptive methods during the study (adequate: combined hormonal contraception associated with inhibition of ovulation, progestogen-only hormonal contraception associated with inhibition of ovulation, intrauterine device, intrauterine hormone-releasing system, bilateral tubal occlusion, vasectomized partner2, sexual abstinence3).

  1. For the purpose of this document, a female is considered of childbearing potential (FCBP), i.e. fertile, following menarche and until becoming post-menopausal unless permanently sterile. Permanent sterilisation methods include hysterectomy, bilateral salpingectomy and bilateral oophorectomy. A postmenopausal state is defined as no menses for 12 months without an alternative medical cause. A high follicle stimulating hormone (FSH) level in the postmenopausal range may be used to confirm a post-menopausal state in women not using hormonal contraception or hormonal replacement therapy. However in the absence of 12 months of amenorrhea, a single FSH measurement is insufficient. For the purpose of this document, a man is considered fertile after puberty unless permanently sterile by bilateral orchidectomy
  2. Vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the WOCBP trial participant and that the vasectomized partner has received medical assessment of the surgical success
  3. In the context of this guidance sexual abstinence is considered a highly effective method only if defined as refraining from heterosexual intercourse during the entire period of risk associated with the study treatments. The reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the subject. 4. All subjects must agree not to share medication. 5. Diagnosis of Idiopathic PD, inclusive of familial PD and genetic forms of L-Dopa responsive PD Age 18 - 75 years 7. Age at Parkinson's disease onset before 65 years 8. Disease duration ≥ 5 years 9. Oral medication constant for four weeks prior to baseline visit 10. Oral treatment with L-Dopa and non-ergot dopamine agonist(s) (any preparation, any dosage) 11. Presence of dopaminergic motor fluctuations based on patient history 12. Presence of dopaminergic neuropsychiatric (affective) fluctuations based on patient history 13. Presence of behavioural hyperdopaminergic syndrome including clinically relevant neuropsychiatric behavioural abnormalities according Ardouin Behavioural Scale Section 1, hypomanic symptoms, psychosis + Section 4 hyperdopaminergic behaviours (score ≥ 3), eventually further accompanied by impulse control disorders, a/o dopamine dysregulation, syndrome, a/o hallucination - psychosis spectrum; in case symptoms of the hallucination/psychosis or hypomania-mania spectrum are present, retained insight is mandatory at the time of study enrolment

Exclusion Criteria:

* 1.Women during pregnancy and lactation. 2. History of hypersensitivity to the investigational medicinal product or to any drug with similar chemical structure or to any excipient present in the pharmaceutical form of the investigational medicinal product. 3. Participation in other clinical trials or observation period of competing trials over the past three months 4. Patients suffering from cognitive impairment (MoCA < 21) will be excluded for the major reason to obtain valid Ardouin assessments that will be hampered in case cognitive impairment (and therefore insight) is too severe 5. Acute paranoid psychosis without retained insight (however impulse control disorder or dopamine dysregulation syndrome are not an exclusion criterion; illusions or (pseudo)-hallucinations are not an exclusion criterion as long as there is no endangerment of the patients themselves or other persons owing to clinical judgement; patients may be eligible after remission of psychosis/suicidality) 6. Severe depression according to ICD-10 criteria; however, affective fluctuations with intermittent depressive symptoms (reversed by dopaminergic medication) are not an exclusion criterion 7. Active suicidality without self-distancing (however, suicidal ideation/thoughts or passive wishes of being dead are not an exclusion criterion as long as the patient is credibly distancing from it). 8. General contraindications for intestinal L-Dopa therapy (according to Lecigon® Fachinformation) 9. Gastrointestinal contraindications against PEG-J tube placement 10. Tremor-dominant PD without dopaminergic response fluctuationt Pre-existing device assisted therapy (DAT) immediately before study enrolment including with DBS, LCIG/LECIG, or subcutaneous therapy with apomorphine or foslevodopa; if patient terminated pre-existing subcutaneous therapy, the patient will be eligible after having received oral dopamine replacement therapy for at least 3 months 12. Malignancy in a non-remitted stage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-16 (Estimated); Primary Completion 2030-09-22 (Estimated); Study Completion 2030-09-22 (Estimated)

PRIMARY OUTCOMES:
Ardouin Behavioral Scale (hyperdopaminergic syndrome) | 6 months
  To show superiority of LECIG therapy compared to best medical treatment on "hyperdopaminergic symptoms" corresponding to Section 1 (items 2 & 4), and section 4 (all items) of the "Ardouin Behavioural Scale" between pre-interventional baseline and 6- month follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Centre for Neurology, Department forNeurodegenerative Disease, and Hertie-Institute forClinical Brain Research, Tübingen, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weintraub D, Koester J, Potenza MN, Siderowf AD, Stacy M, Voon V, Whetteckey J, Wunderlich GR, Lang AE. Impulse control disorders in Parkinson disease: a cross-sectional study of 3090 patients. Arch Neurol. 2010 May;67(5):589-95. doi: 10.1001/archneurol.2010.65. PMID 20457959
- [Background] Lhommee E, Wojtecki L, Czernecki V, Witt K, Maier F, Tonder L, Timmermann L, Halbig TD, Pineau F, Durif F, Witjas T, Pinsker M, Mehdorn M, Sixel-Doring F, Kupsch A, Kruger R, Elben S, Chabardes S, Thobois S, Brefel-Courbon C, Ory-Magne F, Regis JM, Maltete D, Sauvaget A, Rau J, Schnitzler A, Schupbach M, Schade-Brittinger C, Deuschl G, Houeto JL, Krack P; EARLYSTIM study group. Behavioural outcomes of subthalamic stimulation and medical therapy versus medical therapy alone for Parkinson's disease with early motor complications (EARLYSTIM trial): secondary analysis of an open-label randomised trial. Lancet Neurol. 2018 Mar;17(3):223-231. doi: 10.1016/S1474-4422(18)30035-8. PMID 29452685
- [Background] Weintraub D, Mamikonyan E. The Neuropsychiatry of Parkinson Disease: A Perfect Storm. Am J Geriatr Psychiatry. 2019 Sep;27(9):998-1018. doi: 10.1016/j.jagp.2019.03.002. Epub 2019 Mar 9. PMID 31006550
- [Background] Calabresi P, Di Filippo M, Ghiglieri V, Tambasco N, Picconi B. Levodopa-induced dyskinesias in patients with Parkinson's disease: filling the bench-to-bedside gap. Lancet Neurol. 2010 Nov;9(11):1106-17. doi: 10.1016/S1474-4422(10)70218-0. Epub 2010 Sep 27. PMID 20880751
- [Background] Weiss D, Ebersbach G, Moller JC, Schwarz J, Arlt C, Fritz B, Sensken SC, Eggert K. Do we start too late? Insights from the real-world non-interventional BALANCE study on the present use of levodopa/carbidopa intestinal gel in advanced Parkinson's disease in Germany and Switzerland. Parkinsonism Relat Disord. 2022 Oct;103:85-91. doi: 10.1016/j.parkreldis.2022.08.018. Epub 2022 Aug 24. PMID 36087571
- [Background] Weiss D, Jost WH, Szasz JA, Pirtosek Z, Milanov I, Tomantschger V, Kovacs N, Staines H, Amlani B, Smith N, van Laar T. Levodopa-Entacapone-Carbidopa Intrajejunal Infusion in Advanced Parkinson's Disease - Interim Analysis of the ELEGANCE Study. Mov Disord Clin Pract. 2025 Aug;12(8):1075-1085. doi: 10.1002/mdc3.70046. Epub 2025 Mar 25. PMID 40129359
- [Background] Weiss D, Volkmann J, Fasano A, Kuhn A, Krack P, Deuschl G. Changing Gears - DBS For Dopaminergic Desensitization in Parkinson's Disease? Ann Neurol. 2021 Nov;90(5):699-710. doi: 10.1002/ana.26164. Epub 2021 Jul 20. PMID 34235776